CLINICAL TRIAL: NCT06117488
Title: Risk Factors and Management Outcome of Chronic Portal Vein Thrombosis in Children
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Asmaa Aly Fathy Shehata, Principal Investigator, Assiut University
Other Study IDs: chronic portal vein thrombosis
Record Dates: First submitted 2023-10-06; First posted 2023-11-07 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-11

CONDITIONS: Portal Vein Thrombosis
MeSH Terms: interventions — Endoscopy; Dosage Forms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: endoscopy — gastro duodenal endoscoe
  Other Names: drug

SUMMARY:
The aim of study is to evaluate different etiological and risk factors that lead to chronic portal vein thrombosis and to delineate a management plan for chronic portal vein thrombosis in children.

DETAILED DESCRIPTION:
Chronic Portal vein thrombosis (PVT) is deﬁned as thrombosis that develops in the trunk of the portal vein, including its right and/or left intrahepatic branches of more than 5 weeks duration. This thrombus may extend to the splenic or superior mesenteric veins. The causes of chronic PVT in children are not entirely known, but several factors that predispose to this pathology are described. These are classiﬁed into three categories: local factors that can cause injury to the portal vein (abdominal infections, abdominal surgery, umbilical catheter), general factors (procoagulant status), and, less often, vascular malformation. The most common cause is umbilical vein catheterization (UVC). Among the general factors that predispose to venous thrombosis are thrombophilia, sepsis, and dehydration. Deﬁciency or qualitative abnormalities of anti-coagulation factors (antithrombin III, protein C, protein S, and activated protein C resistance) often predispose to thrombotic events, including PVT. Thrombophilia is incriminated in 35% of cases of PVT in children. For this reason, children with PVT, and especially those that associate other risk factors (UVC), should be screened for inherited prothrombotic disorders: prothrombin 20210 mutation (PTHR), factor V Leiden (FVL), methylenetetrahydrofolate reductase (MTHFR) genes deﬁciency, or metabolic defects like hyper homocysteinemia. Congenital abnormalities (portal vein stenosis, atresia, or agenesis) are rarely involved in PVT. Furthermore, early PVT after liver transplantation with cadaveric graft was described in adults. Even less often in children, PVT after splenectomy for hematologic diseases was also described. An association between more than one factor is frequently observed, which further increases the risk of thrombosis. In almost 50% of cases, the etiology of PVT remains unknown.

PVT patients initially present with upper gastrointestinal bleeding (UGIB) or splenomegaly on routine clinical examination in asymptomatic individuals. The initial presence of hematemesis is usually dramatic in a previously healthy child, with past history of morbidity, often without remarkable intercurrent events. Melena may also be observed, but it is less common than hematemesis. The child can be lethargic, with signs of orthostatic hypotension. The clinical examination revealing splenomegaly in a child with UGIB indicates esophageal varices as the most probable site for the bleeding. Less frequently, the diagnosis can be based on the investigation of a child with abdominal pain or with complications related to hypersplenism. The physical examination may reveal splenomegaly; hepatomegaly is not common in children with PVT without underlying liver disease, as well as stigmata of chronic liver disease. PVT should be suspected in all children with splenomegaly, without hepatomegaly and hematemesis, with normal liver function test results. Liver biopsy is normal in children without associated cirrhosis.

Abdominal Doppler ultrasonography is the most widely used diagnostic exam in pediatric patients, with a high sensitivity and specificity, even though it is an operator-dependent diagnostic method. Chronicity of PVT is defined by Doppler ultrasonography by means of visualization of the formation of new vessels around the thrombus (cavernoma). Some diagnostic exams should not be routinely used in pediatric patients due to their risk: splenoportography and arterial portography, nuclear magnetic resonance (angiography), computed tomography (portogram). All patients must be submitted to upper gastrointestinal endoscopy to check for the presence of esophagogastric varices, which will allow for a better planned therapeutic approach. Laboratory exams show normal liver function in most patients, except in those who have a prolonged decrease in portal circulation, or portal biliopathy.

The treatment of portal venous obstruction depends upon the patient's age, the site and nature of the obstruction and the clinical features. Endoscopic variceal ligation (EVL) is the primary choice for the management of variceal bleeding in children. This treatment may be technically difficult in young and small children; sclerotherapy is then recommended as an alternative approach in such cases. Beta adrenergic blockade may play a role in secondary prophylaxis as they reduce the risk of rebleeding and improve survival after variceal bleed. Decompressive shunt surgery should be considered in cases with failed endotherapy. It is also indicated for correcting symptomatic portal hypertensive biliopathy, symptomatic hypersplenism and 'on demand' one-time treatment. Oesophageal transection with or without splenectomy is less useful to control bleeding because of a high risk of late rebleeding and reappearance of varices, but can be resorted to as a nonshunt option in patients with portosystemic encephalopathy, hepatopulmonary syndrome or portopulmonary syndrome. Portal vein thrombosis was considered a major obstacle to liver transplantation which led to increased surgical complexity and perioperative morbidity and mortality.

ELIGIBILITY:
Inclusion Criteria:

- Children and adolescents with Chronic Portal vein thrombosis admitted to Pediatric Gastroenterology, Hepatology and Endoscopy units at Assiut university children hospital (AUCH) in the previous year 2022 from 1/1/2022 to 31/12/2022.

Those with chronic portal vein thrombosis aged from 3 months to 18 years' old.

Exclusion Criteria:

* Patients aged less than 3 months and more than 18 years' old. Those with acute portal vein thrombosis. Children with portal hypertension in absence of chronic portal vein thrombosis.

Ages: 3 Months to 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: Children and adolescents aged from 3 months to 18 years' old. Those with chronic portal vein thrombosis.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2023-11-01 (Estimated); Primary Completion 2024-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Risk Factors and Management Outcome of Chronic Portal Vein Thrombosis in Children | baseline
  -Describe demographic and clinical data of children and adolescents with (PVT) admitted to Pediatric Gastroenterology, Hepatology and Endoscopy units at Assiut university children hospital (AUCH) in the previous year 2022. Assess the outcome of (PVT) in children and adolescents admitted to (AUCH).
  Describe the distribution of etiologies of (PVT) in children and adolescents at Assiut University Children's Hospital.
  -Clinical examination which include:
  * Vital signs: heart rate, blood pressure, respiratory rate, and temperature.
  * General examination: pallor, jaundice and cyanosis.
  * Anthropometric measurements: weight (kg), height (m) and BMI.
  * Cardiac, chest and neurological examination.
  * Local abdominal examination for: abdominal distention, hepatomegaly, splenomegaly, ascites and dilated abdominal wall veins.

CONTACTS AND LOCATIONS:
Overall Officials: Ashraf Mohammed Alsagheer, Lecturer, Study Director — Assiut university, Faculty of midicine